CLINICAL TRIAL: NCT06264050
Title: The Influence of a Psychological Support Group on Mood, Anxiety, Coping Skills of Patients Admitted to Neurorehabilitation: a Pre-post Study
Brief Title: Psychological Support Group and Its Effects on Mood, Anxiety and Coping
Acronym: SUPPORT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Camillo, Venezia, Italy (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023.04
Record Dates: First submitted 2024-02-08; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Coping Strategies; Anxiety; Nurse-Patient Relations; Psychological; Mood Depressed; Rehabilitation; Neurologic Manifestations
MeSH Terms: conditions — Anxiety Disorders; Consciousness Disorders; Neurologic Manifestations

STUDY DESIGN:
Intervention Model Description: pre post study on a single cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients in the psychological support group (Other): Patients in neurorehabilitation attending a psychological support group
  Interventions: Diagnostic Test: evalutaion scales

INTERVENTIONS:
Diagnostic Test: evalutaion scales — four scales will be administered to whom attend a psychological support group: BDI II (depression); Stai Y2 (trait anxiety); Cope NVI 25 (coping strategies) and Core OM (psychological state)

SUMMARY:
The aim of this study is to verify the influence that participation in a Psychological Support Group has on anxiety, depression and coping skills in patients admitted to the IRCCS San Camillo Hospital.

It is therefore an observational study with a pre-post design on a cohort of patients hospitalized at San Camillo IRCCS who attend the Psychological Support Group.

The study consists of verifying whether the therapeutic activity of the Psychological Support Group (GSP) has an influence on the levels of anxiety, mood and coping skills in the patients who attend it. These purposes will be pursued through the administration to each patient at the beginning (pre) and at the end (post) of the period of attendance at the GSP, of validated scales: Stay Y2 (anxiety), BDI II(depressive symptoms), COPE NVD 25 (coping strategies) and the CORE-OM (outcomes of psychological activity).

DETAILED DESCRIPTION:
Several neurological pathologies are associated with a decrease in the quality of life for patients. In particular, previous studies have reported that anxiety and depression are two of the main predictors of this decrease in patients with epilepsy, migraine, multiple sclerosis, Parkinson's disease and stroke. Among these pathologies and in general among the populations of patients with neurological diseases belonging to our hospital, motor, cognitive and communicative impairments negatively impact the quality of life as well as the activities of daily living. Often, these limitations make it necessary to reconceptualise one's personal identity which passes through experiences of acceptance of the disease as well as consolidation of awareness of the disease and of one's functional outcomes (cognitive, motor, etc.) with consequent repercussions in terms of the tone of the mood such as experiences of anxiety and depression.

A psychological support intervention is therefore necessary, after evaluating these aspects, in order to outline the critical issues as well as the possible compensation factors that can be provided to the patient in order to strengthen his motivation for the treatment and in general for the rehabilitation process during the hospitalization period, favoring the emergence of more functional coping strategies. Often, in fact, the patient is not able to ask for support or help from operators and/or family members, is not able to appropriately manage their emotional experiences and often experiences incongruent feelings of guilt. These aspects negatively influence the rehabilitation services received and generally outline a hospitalization experience that is not entirely functional. From this perspective, in addition to the individual psychological path, the possibility of accessing a psychological support group is configured as a suitable treatment space-time in which to express one's needs and concerns for the future, where issues relating to the condition can be explored in depth. existential. This is undoubtedly the starting point: the desire to understand, the desire to understand the disease, but also the expectations and fears in order to understand the disease and implement more realistic and congruent expectations in view of relational and professional reintegration, where possible .

The aim of this study is to verify what influence attending the Psychological Support Group has on anxiety, depressive symptoms, coping styles and what psychological outcomes it leads to in neurorehabilitation patients.

Outcomes:

For the STAI Y2 Scale, a score lower than 50 is indicative of a decrease in state anxiety.

For the BDI II, an improvement in depressive symptoms is expected which will be expressed with a change in score range (for example from moderate to light, i.e. going from the range 20-28 to 14-19) or with a decrease in the score within the same range (for example in the severe range).

For the CORE OM, the total raw scores (0-136) of the entire scale will be analysed, also adding the scores of the 4 individual dimensions. It is expected that the score at the second post survey will decrease both in the general sum of the 34 items and in the individual dimensions.

Subsequently, the correlations between the factors will be searched for and analyzed with the Pearson r coefficient.For the COPE NVI 25 Scale, the scores of the individual dimensions will be added and given that a higher score corresponds to a better predisposition, it is expected that the dimensions "Orientation to the problem" will increase, "Positive attitude" will increase, "Transcendent orientation" will increase, so such as "Social support" while "Avoidance strategies" decreases in the score.

Subsequently, the correlations between the factors will be searched for and analyzed with the Pearson r coefficient.

Sample:

Patients undergoing neurorehabilitation admitted to the IRCCS San Camillo for whom there is an indication of participation in the Psychological Support Group held by the Neuropsychology Service of the IRCCS San Camillo will be considered eligible for the study.

Procedure The patient who receives the indication to be part of the Psychological Support Group and who meets the inclusion and exclusion criteria will be contacted by a researcher who, after obtaining consent, the day before starting participation in the GSP, will ask the patient the rating scales will be administered (pre - T1 phase). We assume around 30 minutes to compile When the patient finishes participating in the support group, the researcher/interviewer will repeat the administration of the same scales, according to the methods and precautions described above (post-T2 phase) the day after discharge from the GSP.

The scales will be administered and carried out by specially trained psychological and nursing staff who will not correspond with the staff who will conduct the GSP. Patient data will be anonymized.

The following information and data will be collected from clinical documentation.

* Gender, age, educational qualification, current profession or before retirement, marital status, presence of children or social network
* Main pathology (cause of entry into neurorehabilitation) and types of main pathology (e.g. type of stroke and its location), main comorbidities.
* Duration of hospitalization at T0, duration of the pathology, number of hospitalizations (whether first hospitalization or not).
* Barthel Index and FIM (Functional Independence Measure) scale, both at T0 and T2 These two scales are already present in the medical record because they are a routine and mandatory part of hospitalization In addition to the descriptive statistics, the Student's t test for paired data will be applied, or the non-parametric equivalent (Wilcoxon signed-rank test). The normality of the variables will be tested using the Shapiro-Wilk test.

Two-tailed tests with an alpha error of 0.05 will be used. The collected data will be processed using STATA software (version 15 or higher).

The sample size was calculated on the BDI-II scale due to its clinical relevance in neurorehabilitation treatment (Wang & Gorestain, 2013). Given the scarcity of studies in patients undergoing neurorehabilitation, the standard deviation reported by Huang et al (2017) on a sample of patients with Parkinson's disease equal to 8.4 was used.

Assuming a clinically relevant mean difference in the raw scores of 6 (effect size 0.71), 19 subjects will be necessary, considering a two-tailed test, a type I error of 5% and a power of 80%. Taking into account a possible dropout rate of 20%, the subjects to be enrolled become 24. The calculation was carried out using the G-Power software (version 3.1.9.6) using the Wilcoxon signed-rank test (for difference in average for paired data).

Expected results:

Patients who attend the Psychological Support Group are expected to have a general improvement in their psychological condition related to hospitalization and illness. Reduction in anxiety levels, fewer depressive symptoms and development of more effective coping strategies.

ELIGIBILITY:
Inclusion Criteria:

Patients hospitalized at the IRCCS San Camillo. Patients with indication to attend the Psychological Support Group. Patients who have given valid consent. Patients able to understand and read Italian. Patients with any type of neurological pathology for which they are admitted to neurorehabilitation.

Aphasic patients without comprehension deficits and able to communicate effectively with augmented communication media.

Exclusion Criteria:

Patients unable to give valid consent. Minor patients or patients over 85 years of age. Patients with participation in the Psychological Support Group of less than three sessions.

Patients with cognitive deficits that prevent them from completing the scales and taking the interview.

Patients unable to understand and read Italian. Patients with pathologies for which they are not undergoing neurorehabilitation treatment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2004-01-08 (Actual); Primary Completion 2024-09-08 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
The State-Trait Anxiety Inventory (STAI) Y2 | 10 minutes
  The Stai Y2 instead measures state anxiety (State-anxiety), i.e. a transitory emotional state of an individual in a particular situation, unlike trait anxiety (Trait-anxiety) which reflects a personality variable that stably characterizes the individual and differentiates him from others in the propensity to respond with high levels of anxiety to situations perceived as dangerous. Trait anxiety is measured by the Stai version Y1
The Beck Depression Inventory II (BDI-II) | 15 minutes
  The Beck Depression Inventory II (BDI-II) has 21 items on a 4-point Likert scale (from 0 to 3) and a total score ranging from 0 to 63. Given that the BDI does not diagnose depression but the presence of depressive symptoms, according the manual scores from 0 to 13 indicate normality, from 14 to 19 mild depression, from 20 to 28 moderate depression, from 29 to 63 severe depression.
The Clinical Outcomes in Routine Evaluation-Outcome Measure (CORE-OM) | 20 minutes
  The Clinical Outcomes in Routine Evaluation-Outcome Measure (CORE-OM) is a 34-item self-report instrument for measuring outcomes in psychological treatments that has been shown to be reliable, valid, and acceptable in various clinical settings. The items cover four domains: subjective well-being, problems/symptoms, life functioning, and risk. Higher scores in all domains indicate greater psychological problems
The Coping Orientations to Problem Experienced NVI - 25 | 15 minutes
  The Coping Orientations to Problem Experienced is a self-report questionnaire that takes into consideration different coping methods. The questionnaire asks you to evaluate how often the subject implements that particular coping process in difficult or stressful situations; There are four answer possibilities, from "I usually don't do it" to "I almost always do it". The short version validated in Italian (NVI) has 25 items instead of the 60 of the original version.
  All elements were grouped into 5 subdimensions, namely: Avoidance strategies, Transcendental orientation, Positive attitude, Social support, Problem orientation.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Camuccio, doctor, Principal Investigator — IRCCS San Camillo

REFERENCES:
- [Result] Castelnuovo G, Giusti EM, Manzoni GM, Saviola D, Gatti A, Gabrielli S, Lacerenza M, Pietrabissa G, Cattivelli R, Spatola CA, Corti S, Novelli M, Villa V, Cottini A, Lai C, Pagnini F, Castelli L, Tavola M, Torta R, Arreghini M, Zanini L, Brunani A, Capodaglio P, D'Aniello GE, Scarpina F, Brioschi A, Priano L, Mauro A, Riva G, Repetto C, Regalia C, Molinari E, Notaro P, Paolucci S, Sandrini G, Simpson SG, Wiederhold B, Tamburin S. Psychological Treatments and Psychotherapies in the Neurorehabilitation of Pain: Evidences and Recommendations from the Italian Consensus Conference on Pain in Neurorehabilitation. Front Psychol. 2016 Feb 19;7:115. doi: 10.3389/fpsyg.2016.00115. eCollection 2016. PMID 26924998
- [Result] Chiu EC, Chen YJ, Wu WC, Chou CX, Yu MY. Psychometric Comparisons of Three Depression Measures for Patients With Stroke. Am J Occup Ther. 2022 Jul 1;76(4):7604205140. doi: 10.5014/ajot.2022.049347. PMID 35727642
- [Result] Denham AMJ, Baker AL, Spratt N, Guillaumier A, Wynne O, Turner A, Magin P, Bonevski B. The unmet needs of informal carers of stroke survivors: a protocol for a systematic review of quantitative and qualitative studies. BMJ Open. 2018 Jan 31;8(1):e019571. doi: 10.1136/bmjopen-2017-019571. PMID 29391371
- [Result] Gregorio GW, Brands I, Stapert S, Verhey FR, van Heugten CM. Assessments of coping after acquired brain injury: a systematic review of instrument conceptualization, feasibility, and psychometric properties. J Head Trauma Rehabil. 2014 May-Jun;29(3):E30-42. doi: 10.1097/HTR.0b013e31828f93db. PMID 23640542
- [Result] Huang SL, Hsieh CL, Wu RM, Lu WS. Test-retest reliability and minimal detectable change of the Beck Depression Inventory and the Taiwan Geriatric Depression Scale in patients with Parkinson's disease. PLoS One. 2017 Sep 25;12(9):e0184823. doi: 10.1371/journal.pone.0184823. eCollection 2017. PMID 28945776
- [Result] Kampling H, Reese C, Kust J, Mittag O. Systematic development of practice guidelines for psychological interventions in stroke rehabilitation. Disabil Rehabil. 2020 Jun;42(11):1616-1622. doi: 10.1080/09638288.2018.1530308. Epub 2019 Jan 7. PMID 30616425
- [Result] Liao B, Liang M, Ouyang Q, Song H, Chen X, Su Y. Psychological Nursing of Patients With Stroke in China: A Systematic Review and Meta-Analysis. Front Psychiatry. 2020 Dec 11;11:569426. doi: 10.3389/fpsyt.2020.569426. eCollection 2020. PMID 33362596
- [Result] Palmieri G, Evans C, Hansen V, Brancaleoni G, Ferrari S, Porcelli P, Reitano F, Rigatelli M. Validation of the Italian version of the Clinical Outcomes in Routine Evaluation Outcome Measure (CORE-OM). Clin Psychol Psychother. 2009 Sep-Oct;16(5):444-9. doi: 10.1002/cpp.646. PMID 19701881
- [Result] Pearce G, Pinnock H, Epiphaniou E, Parke HL, Heavey E, Griffiths CJ, Greenhalgh T, Sheikh A, Taylor SJ. Experiences of Self-Management Support Following a Stroke: A Meta-Review of Qualitative Systematic Reviews. PLoS One. 2015 Dec 14;10(12):e0141803. doi: 10.1371/journal.pone.0141803. eCollection 2015. PMID 26657458
- [Result] Raciti L, Corallo F, Manuli A, Calabro RS. Nursing, Caregiving and Psychological support in Chronic Disorders of Consciousness: a scoping review. Acta Biomed. 2021 Mar 31;92(S2):e2021013. doi: 10.23750/abm.v92iS2.11329. PMID 33855992
- [Result] Santangelo G, Sacco R, Siciliano M, Bisecco A, Muzzo G, Docimo R, De Stefano M, Bonavita S, Lavorgna L, Tedeschi G, Trojano L, Gallo A. Anxiety in Multiple Sclerosis: psychometric properties of the State-Trait Anxiety Inventory. Acta Neurol Scand. 2016 Dec;134(6):458-466. doi: 10.1111/ane.12564. Epub 2016 Feb 1. PMID 27219913
- [Result] Sarkamo T. Cognitive, emotional, and neural benefits of musical leisure activities in aging and neurological rehabilitation: A critical review. Ann Phys Rehabil Med. 2018 Nov;61(6):414-418. doi: 10.1016/j.rehab.2017.03.006. Epub 2017 Apr 29. PMID 28461128
- [Result] Sihvonen AJ, Sarkamo T, Leo V, Tervaniemi M, Altenmuller E, Soinila S. Music-based interventions in neurological rehabilitation. Lancet Neurol. 2017 Aug;16(8):648-660. doi: 10.1016/S1474-4422(17)30168-0. Epub 2017 Jun 26. PMID 28663005
- [Result] Soratto J, Pires DEP, Friese S. Thematic content analysis using ATLAS.ti software: Potentialities for researchs in health. Rev Bras Enferm. 2020 Apr 22;73(3):e20190250. doi: 10.1590/0034-7167-2019-0250. eCollection 2020. PMID 32321144
- [Result] Starkstein SE, Lischinsky A. The phenomenology of depression after brain injury. NeuroRehabilitation. 2002;17(2):105-13. PMID 12082237
- [Result] Wang YP, Gorenstein C. Assessment of depression in medical patients: a systematic review of the utility of the Beck Depression Inventory-II. Clinics (Sao Paulo). 2013 Sep;68(9):1274-87. doi: 10.6061/clinics/2013(09)15. PMID 24141845